CLINICAL TRIAL: NCT01377493
Title: Effects of a Chewing Gum Containing POs-Ca and Fluoride on Remineralization of Enamel Subsurface Lesions in Situ
Brief Title: Effects of a Chewing Gum Containing POs-Ca and Fluoride on Enamel
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Tokyo Medical and Dental University (Other)
Responsible Party: Yuichi Kitasako, Tokyo Medical and Dental University
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: 1B116
Record Dates: First submitted 2011-06-17; First posted 2011-06-21 (Estimated); Last update posted 2011-06-21 (Estimated); Status verified 2011-06

CONDITIONS: Enamel Subsurface Lesion
Keywords: chewing-gum; enamel subsurface lesion; calcium additives; fluoride; in situ
MeSH Terms: interventions — Chewing Gum

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- placebo (Placebo Comparator)
  Interventions: Dietary Supplement: chewing gum
- POs-Ca (Active Comparator)
  Interventions: Dietary Supplement: chewing gum
- POs-Ca+F (Active Comparator)
  Interventions: Dietary Supplement: chewing gum

INTERVENTIONS:
Dietary Supplement: chewing gum — chewing gum containing no active ingredients, or Ca-P bioavailable ions, or Ca-P and F bioavailable ions

SUMMARY:
There were no differences in the degree of enamel remineralization of subsurface lesions among the chewing gums containing or not containing POs-Ca and fluoride.

ELIGIBILITY:
Inclusion Criteria:

* healthy adult subjects
* More than 22 permanent teeth

Exclusion Criteria:

* Alcohol addiction
* Smoking
* Active caries
* Periodontal pockets
* Low-saliva flow (less than 0.3ml/min)

Ages: 20 Years to 31 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 36 (Actual)
Dates: Start 2009-12; Primary Completion 2010-02 (Actual); Study Completion 2011-06 (Actual)

PRIMARY OUTCOMES:
Mineral content of enamel | 2 weeks
  Mineral content of bovine enamel blocks inserted into the subject mouth during chewing of the gums was assessed.

REFERENCES:
- [Derived] Kitasako Y, Sadr A, Hamba H, Ikeda M, Tagami J. Gum containing calcium fluoride reinforces enamel subsurface lesions in situ. J Dent Res. 2012 Apr;91(4):370-5. doi: 10.1177/0022034512439716. Epub 2012 Feb 15. PMID 22337700
- [Derived] Kitasako Y, Tanaka M, Sadr A, Hamba H, Ikeda M, Tagami J. Effects of a chewing gum containing phosphoryl oligosaccharides of calcium (POs-Ca) and fluoride on remineralization and crystallization of enamel subsurface lesions in situ. J Dent. 2011 Nov;39(11):771-9. doi: 10.1016/j.jdent.2011.08.009. Epub 2011 Aug 19. PMID 21875640